CLINICAL TRIAL: NCT00355888
Title: A Phase I, Open Label Study of MBP-426 Given by Intravenous Infusion in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Safety Study of MBP-426 (Liposomal Oxaliplatin Suspension for Injection) to Treat Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mebiopharm Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M05-10070
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2009-09

CONDITIONS: Cancer
Keywords: Cancer; Advanced or Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label study of MBP-426 (Experimental): Dose escalation starting at 6 mg/m2, IV (in the vein) on Day 1 of each 21-day cycle. Number of Cycles: Up to 6 cycles, until unacceptable toxicity, disease progression, or intercurrent illness requires treatment discontinuation. Patients may continue treatment beyond 6 cycles if the Investigator determines that additional treatment would provide further benefit for the patient as long as toxicity remains acceptable.
  Interventions: Drug: MBP-426

INTERVENTIONS:
Drug: MBP-426 — Dose escalation starting at 6 mg/m2, IV (in the vein) on Day 1 of each 21-day cycle. Number of Cycles: Up to 6 cycles, until unacceptable toxicity, disease progression, or intercurrent illness requires treatment discontinuation. Patients may continue treatment beyond 6 cycles if the Investigator determines that additional treatment would provide further benefit for the patient as long as toxicity remains acceptable.

SUMMARY:
The purpose of this study is to determine whether MBP-426 (liposomal oxaliplatin suspension for injection) is safe and effective in the treatment of advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Study Phase 1 Study Type (Interventional/Observational) Interventional Study Design Purpose: Treatment Allocation: Nonrandomized trial Masking: Open Control: Dose Comparison Assignment: Single Group Endpoint: Safety/Efficacy

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed malignancy that is locally advanced or metastatic solid tumor and is refractory to standard therapy or for which conventional therapy is not reliably effective or no effective therapy is available
* 18 years of age or older
* ECOG Performance Status of 0, 1, or 2
* Adequate clinical laboratory values:

  * absolute neutrophil count greater than or equal to 1500 cells/microliter
  * platelets greater than or equal to 100,000 cells/microliter
  * serum creatinine less than or equal to 1.5 x upper limit of normal (ULN) for the institution
  * creatinine clearance (calculated) > 60 mL/min (using the Cockcroft-Gault equation)
  * bilirubin less than or equal to 1.5 x ULN
  * alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 2.5 x ULN (patients with known liver metastases may have up to 5 times ULN AST and ALT levels).
* Ability to cooperate with treatment and follow-up schedules
* Negative pregnancy test and using at least one form of contraception as approved by the Investigator prior to study entry if a female patient of childbearing potential or a male patient with a female partner of childbearing potential
* Measurable disease as defined by RECIST criteria or non-measurable disease
* Patients with known brain metastases may be included as long as they have been clinically stable for one month or more, and are not receiving dexamethasone
* Ability to maintain a central intravenous access (e.g. PICC, Groshong, or Hickman line)
* Signed informed consent prior to the start of any study specific procedures

Exclusion Criteria:

* Received previous anticancer chemotherapy, immunotherapy, radiotherapy or any other investigational therapy in the 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study entry
* Received extensive prior radiotherapy to more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation
* Any concomitant condition that could compromise the objectives of this study and the patient's compliance
* Pregnant or lactating women
* Current malignancies of another type, with the exception of adequately treated in situ cervical cancer and basal cell skin cancer or have demonstrated no evidence of disease for 5 years or more
* Clinically evident HIV, HBV, or HCV infection
* Hematologic malignancy
* Documented or known bleeding disorder
* Requirements for therapeutic anticoagulation that increases INR or aPTT above the normal range (low dose deep vein thrombosis [DVT] or line prophylaxis is allowed)
* Congestive heart failure
* Greater than Grade 1 peripheral neuropathy according to the National Cancer Institute's Common Terminology Criteria for Adverse Events v3.0 (CTCAE version 3.0)
* History of allergic reactions to platinum-based or liposomal agents
* Creatinine clearance (calculated) less than or equal to 60 mL/min (using the Cockcroft-Gault equation)
* Receiving or initiating treatment with any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-06; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity, determination of maximum tolerated dose (MTD), and recommended Phase 2 dose | Within 21 days of treatment administration

SECONDARY OUTCOMES:
Tumor shrinkage according to RECIST | Measured every 6 weeks (i.e., every 2 cycles) while receiving study drug
Limited exploratory assays | Variable throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Alexandria Phan, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - M.D. Anderson Cancer Center, Houston, Texas
  - Institute for Drug Development, San Antonio, Texas

REFERENCES:
- [Derived] Alavi N, Rezaei M, Maghami P, Fanipakdel A, Avan A. Nanocarrier System for Increasing the Therapeutic Efficacy of Oxaliplatin. Curr Cancer Drug Targets. 2022;22(5):361-372. doi: 10.2174/1568009622666220120115140. PMID 35048809